CLINICAL TRIAL: NCT04528277
Title: Role of Short Course Rifapentine and Isoniazid for the Preventive Treatment for Latent Genital Tuberculosis in Women With Recurrent Implantation Failure: A Prospective Interventional Cohort Study
Brief Title: Short Course Rifapentine and Isoniazid for the Preventive Treatment for Latent Genital Tuberculosis
Acronym: SCRIPT-LGTB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, director of department of infectious diseases, Huashan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KS20232
Record Dates: First submitted 2020-08-22; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Infertility, Female; Recurrent Implantation Failure; Genital Tuberculoses, Female; Genital Tuberculosis, Latent
MeSH Terms: conditions — Infertility, Female; Tuberculosis, Female Genital | interventions — rifapentine; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- LGTB treatment group (Experimental): The LGTB treatment group will receive the 1-month regimen of three times weekly rifapentine (150mg per capsule, 450mg po tiw) plus isoniazid (100mg per tablet, 400mg po tiw).
  Interventions: Drug: rifapentine plus isoniazid
- LGTB no treatment group (No Intervention): The LGTB no treatment group will not take any medication related to preventive treatment of tuberculosis.
- non-LGTB group (No Intervention): The non-LGTB group will not take any medication related to preventive treatment of tuberculosis.

INTERVENTIONS:
Drug: rifapentine plus isoniazid — receive the 1-month regimen of three times weekly rifapentine (450mg po) plus isoniazid (400mg po)
  Arms: LGTB treatment group

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of the 1-month regimen of three times weekly rifapentine plus isoniazid in improving fertility outcome in recurrent implantation failure (RIF) patients with latent genital tuberculosis (LGTB), compared to no treatment and non-LGTB patients.

DETAILED DESCRIPTION:
The prevalence of latent genital tuberculosis (LGTB) is relatively high in women with infertility and recurrent pregnancy loss. Whether preventive treatment of latent tuberculosis infection (LTBI) can improve the fertility outcome in women with recurrent implantation failure (RIF) remains to be explored.

This is a prospective interventional cohort study.The main purpose of this study is to compare the fertility outcome between 1-month regimen of three times weekly rifapentine plus isoniazid and no treatment in RIF patients with LGTB and RIF patients without LGTB. The study will also assess the safety and tolerability and the efficacy of the preventive treatment regimen in prevention of the incidence of active female genital tuberculosis (FGTB).

A total of 1050 participants will be recruited for screening of LGTB. The endometrial tuberculosis (TB) polymerase chain reaction (PCR) test will be employed for the diagnosis of LGTB. Eligible participants with negative TB PCR results will be assigned to the non-LGTB group, while those with positive TB PCR results will be assigned to the LGTB group. The LGTB group will be further assigned, according to their will to receive preventive treatment of tuberculosis, to one of the following groups: the LGTB treatment group and the LGTB no treatment group.

The LGTB treatment group will receive the 1-month regimen of three times weekly rifapentine plus isoniazid, and the in vitro fertilization (IVF)/ intra cytoplasmic sperm injection (ICSI) cycle can be started after 1 month post the completion of the treatment regimen. Adverse events and side effects will be monitored at a 2-week interval during the preventive treatment and followed up once more at 4 weeks post the end of treatment. The LGTB no treatment group and the non-LGTB group will start the IVF/ICSI cycle directly after enrollment without taking any medication related to preventive treatment of tuberculosis.

Eligible participants will be followed up until the end of an IVF/ ICSI cycle or pregnancy. Fertility outcomes of both groups will be recorded and compared. Secondary outcomes, including the incidence of adverse events, the adhesion of treatment and the incidence of LGTB and FGTB, ovarian reserve, embryo quality, history of infertility and tuberculosis will also be recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 25-40 years old
2. Infertile women failed to achieve clinical pregnancy after 4 good quality embryo transfers, with at least 3 fresh or frozen IVF cycles
3. Intended to undergo IVF/ICSI
4. Ultrasonography or hysterosalpingogram showed a normal uterus cavity, and the thickness of the endometrium was ≥8mm before implantation during last IVF/ICSI cycle
5. Patients who voluntarily signed the informed consent and agreed to be followed up as required by the study protocol

Exclusion Criteria:

1. Use of donor eggs/sperm
2. An abnormal uterine cavity shown on hysterosalpingogram or hysteroscopy
3. Proven tubal infertility
4. Proven preimplantation genetic abnormality
5. Proven active tuberculosis
6. Treated for active tuberculosis or used preventive treatment for LTBI within 2 years
7. Being allergic or intolerant of any study drug
8. HIV antibody positive and AIDS patients
9. Patients with impaired liver function: hepatic encephalopathy, ascites; total bilirubin is more than 2 times higher than the upper limit of normal; alanine transaminase (ALT) or aspartate aminotransferase (AST) is more than 5 times the upper limit of normal
10. Patients with diabetes mellitus
11. Critically ill patients, and according to the judgment of the research physician, it is impossible to survive for more than 16 weeks
12. Currently participating in another drug clinical trial

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1050 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rates | 6 weeks after completion of an IVF/ICSI cycle
  Clinical pregnancy was defined as the presence of at least one gestational sac on ultrasound at 6 weeks.
Ongoing Pregnancy Rate | 10 weeks after completion of an IVF/ICSI cycle
  Ongoing pregnancy was the presence of at least one foetus with heart pulsation on ultrasound beyond 10 weeks.
Miscarriage rate | 22 weeks after completion of an IVF/ICSI cycle
  The number of miscarriages before 22 weeks divided by the number of participants with positive pregnancy test.

SECONDARY OUTCOMES:
Implantation rate | 6 weeks after completion of an IVF/ICSI cycle
  The number of gestational sacs seen on scanning divided by the number of embryos replaced.
Incidence of LGTB | 4 weeks after enrollment
  The number of participants diagnosed with LGTB devided by the number of participants screened for LGTB.
Incidence of FGTB | 2 years
  The number of participants developed FGTB during treatment or follow-up devided by the number of participants in the LGTB treatment group.
Incidence of grade 3 or greater adverse events | 20 weeks after preventive treatment initiated
  The number of participants reported grade 3 or greater adverse events during treatment or follow-up devided by the number of participants in the LGTB treatment group.
Completion rate of preventive treatment | 20 weeks after preventive treatment initiated
  11 or 12 doses of the 1-month preventive treatment regimen of three times weekly rifapentine plus isoniazid taken within 16 weeks after treatment initiated will be regarded as completion of preventive treatment. The number of participants completed treatment devided by the number of participants initiated the preventive treatment.
Discontinuation of treatment | 20 weeks after preventive treatment initiated
  The number of participants discontinued treatment devided by the number of participants in the LGTB treatment group.
Discontinuation of treatment due to side effect of study drugs | 20 weeks after preventive treatment initiated
  The number of participants discontinued treatment due to side effect of study drugs devided by the number of participants in the LGTB treatment group.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grace GA, Devaleenal DB, Natrajan M. Genital tuberculosis in females. Indian J Med Res. 2017 Apr;145(4):425-436. doi: 10.4103/ijmr.IJMR_1550_15. PMID 28862174
- [Background] Jindal UN, Verma S, Bala Y. Favorable infertility outcomes following anti-tubercular treatment prescribed on the sole basis of a positive polymerase chain reaction test for endometrial tuberculosis. Hum Reprod. 2012 May;27(5):1368-74. doi: 10.1093/humrep/des076. Epub 2012 Mar 14. PMID 22419745
- [Background] Dam P, Shirazee HH, Goswami SK, Ghosh S, Ganesh A, Chaudhury K, Chakravarty B. Role of latent genital tuberculosis in repeated IVF failure in the Indian clinical setting. Gynecol Obstet Invest. 2006;61(4):223-7. doi: 10.1159/000091498. Epub 2006 Feb 13. PMID 16479141
- [Background] Jirge PR, Chougule SM, Keni A, Kumar S, Modi D. Latent genital tuberculosis adversely affects the ovarian reserve in infertile women. Hum Reprod. 2018 Jul 1;33(7):1262-1269. doi: 10.1093/humrep/dey117. PMID 29897442
- [Background] Bagchi B, Chatterjee S, Gon Chowdhury R. Role of latent female genital tuberculosis in recurrent early pregnancy loss: A retrospective analysis. Int J Reprod Biomed. 2019 Dec 30;17(12):929-934. doi: 10.18502/ijrm.v17i12.5799. eCollection 2019 Dec. PMID 32095740